CLINICAL TRIAL: NCT02902614
Title: Effect of Embryo Biopsy Side on Post Biopsy Blastocyst Structurs and Implantation
Brief Title: Side of Embryo Biopsy Interfering Implantation Potential
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmad Mustafa Mohamed Metwalley (Other)
Collaborators: Ibn Sina Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Ahmad Mustafa Mohamed Metwalley, IVF laboratory manager, Al Baraka Fertility Hospital
Organization: Al Baraka Fertility Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Embryo Biopsy
Record Dates: First submitted 2016-09-07; First posted 2016-09-16 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Preimplantation Diagnosis
Keywords: embryo biopsy; preimplantation genetic testing; animal pole; vegetal pole; day 3 embryo biopsy; embryo implantation; Blastomeres

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vegetal Pole blastomer embryo (Experimental): for day 3 embryo biopsy / cleavage stage: Blastomere collection from opposite side to the 2nd polar body or from vegetal pole.
  Interventions: Procedure: Vegetal Pole blastomer embryo; Procedure: Animal Pole blastomer embryo
- Animal Pole blastomer embryo (Experimental): for day 3 embryo biopsy / cleavage stage: Blastomere collection from and side around the 2nd polar body and not the vegetal pole.
  Interventions: Procedure: Vegetal Pole blastomer embryo; Procedure: Animal Pole blastomer embryo

INTERVENTIONS:
Procedure: Vegetal Pole blastomer embryo — for day 3 embryo biopsy / cleavage stage
  Other Names: Biopsy embryo from sides considered far from ICM location.
Procedure: Animal Pole blastomer embryo — for day 3 embryo biopsy / cleavage stage
  Other Names: Random biopsy without considering specific location

SUMMARY:
Selection of side of embryo biopsy that will not interfering with implantation power of developed blastocyst embryo during biopsy procedure arranged for PGT.

DETAILED DESCRIPTION:
During process of embryo biopsy, it was indicated to avoid contacting cells closer to inner cell mass as it can decrease the quality of embryo and its structural composition. However, recommendation for collection from the trophectoderm (TE) side is indicated.

Absence of differentiation during cleavage-stage or morula stage at day 3 and day 4 respectively, will present the needful to focus a specific location for embryo biopsy during pre-blastocyst stages for embryo going to do genetic testing before implantation or embryo transfer.

In articulation around the second polar body or the animal pole of embryo, collection of the cell from the vegetal pole in crospondence to avoide collection form the animal pole is to be compare the results of implantation for biopsy done using the animal pole side or the random non organized biosy procedure.

ELIGIBILITY:
Inclusion Criteria:

* grade 1 or 2 embryos at eight cell stage or 8-1/ 8-2 embryo quality.

Exclusion Criteria:

* grade 3 embryo at day 3, or 8-3 embryos.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-02 (Actual)

PRIMARY OUTCOMES:
blastocyst location of ICM at day 5 | 2 months
  describing the location of the inner cell mass (ICM) in location to the zona peluceda (ZP) drilling opening.

SECONDARY OUTCOMES:
Implantation power | 2 months
  calculating the pregnancy rate for cases after biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M Metwalley, Principal Investigator — Al Baraka Fertility Hospital
Locations (2):
- AHMAD Barakat, Manama, Bahrain
- Ibn Sina IVF Center- Ibn Sina Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After abstract submission or after final approval for scientific paper

REFERENCES:
- [Result] Tscherne RJ, Capitano G. High-pressure liquid chromatographic separation of pharmaceutical compounds using a mobile phase containing silver nitrate. J Chromatogr. 1977 Jun 11;136(2):337-41. doi: 10.1016/s0021-9673(00)86290-1. No abstract available. PMID 195970
- [Result] Geraedts J, Sermon K. Preimplantation genetic screening 2.0: the theory. Mol Hum Reprod. 2016 Aug;22(8):839-44. doi: 10.1093/molehr/gaw033. Epub 2016 Jun 2. PMID 27256482
- [Result] Balakier H, Sojecki A, Motamedi G, Librach C. Impact of multinucleated blastomeres on embryo developmental competence, morphokinetics, and aneuploidy. Fertil Steril. 2016 Sep 1;106(3):608-614.e2. doi: 10.1016/j.fertnstert.2016.04.041. Epub 2016 May 18. PMID 27206619
- [Result] Cimadomo D, Capalbo A, Ubaldi FM, Scarica C, Palagiano A, Canipari R, Rienzi L. The Impact of Biopsy on Human Embryo Developmental Potential during Preimplantation Genetic Diagnosis. Biomed Res Int. 2016;2016:7193075. doi: 10.1155/2016/7193075. Epub 2016 Jan 28. PMID 26942198
- [Result] Wang Z, Ang WT, Tan SY, Latt WT. Automatic segmentation of zona pellucida and its application in cleavage-stage embryo biopsy position selection. Annu Int Conf IEEE Eng Med Biol Soc. 2015;2015:3859-64. doi: 10.1109/EMBC.2015.7319236. PMID 26737136
- [Result] Dahdouh EM, Balayla J, Audibert F; Genetics Committee; Wilson RD, Audibert F, Brock JA, Campagnolo C, Carroll J, Chong K, Gagnon A, Johnson JA, MacDonald W, Okun N, Pastuck M, Vallee-Pouliot K. RETIRED: Technical Update: Preimplantation Genetic Diagnosis and Screening. J Obstet Gynaecol Can. 2015 May;37(5):451-63. doi: 10.1016/s1701-2163(15)30261-9. PMID 26168107
- See also: Oct4 and Sox2 Directly Regulate Expression of Another Pluripotency Transcription Factor, Zfp206, in Embryonic Stem Cells — http://www.jbc.org/content/282/17/12822.full
- See also: Oct4/Sox2 Binding Sites Contribute to Maintaining Hypomethylation of the Maternal Igf2/H19 Imprinting Control Region — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0081962
- See also: Formation of Pluripotent Stem Cells in the Mammalian Embryo Depends on the POU Transcription Factor Oct4 — http://dx.doi.org/10.1016/S0092-8674(00)81769-9
- See also: Multipotent cell lineages in early mouse development depend on SOX2 function — http://www.ncbi.nlm.nih.gov/pubmed/12514105